CLINICAL TRIAL: NCT03821467
Title: Short- and Long-term Reproducibility of Dual Beam Doppler Fourier-domain Optical Coherence Tomography Measurements in Healthy Subjects - a Pilot Study
Brief Title: Reproducibility of Dual Beam Doppler Fourier-domain Optical Coherence Tomography in Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Associate Professor, MD, PhD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-010418
Record Dates: First submitted 2019-01-28; First posted 2019-01-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Ocular Blood Flow
Keywords: doppler optical coherence tomography; dynamic vessel analyzer
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy subjects (Experimental): Dual beam Doppler Fourier-domain OCT (DOCT) Dynamic Vessel Analyzer (DVA) Optical coherence tomography (OCT)
  Interventions: Device: Dual beam Doppler Fourier-domain OCT (DOCT); Device: Dynamic Vessel Analyzer (DVA); Device: Optical coherence tomography (OCT)

INTERVENTIONS:
Device: Dual beam Doppler Fourier-domain OCT (DOCT) — Retinal blood flow will be assessed using DOCT.
Device: Dynamic Vessel Analyzer (DVA) — Retinal vessel diameters and oxygen saturation will be measured with the DVA device.
Device: Optical coherence tomography (OCT) — Retinal morphology will be imaged using OCT.

SUMMARY:
Dual beam Doppler Fourier-domain Optical coherence tomography (DOCT) is a noninvasive technique to quantify total retinal blood flow.

To enable further development of this technique it is essential to assess short- and long-term reproducibility of DOCT blood flow measurements.

DETAILED DESCRIPTION:
In the present study, total retinal blood flow will be measured with DOCT at multiple time points to gain information of short- and long-term reproducibility. In addition, provocation with flickering light will be performed, which is known to lead to vasodilatation and an increase in retinal blood flow in healthy subjects. Vessel diameters will also be measured using the Dynamic Vessel Analyzer (DVA).

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years
* Non-smokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropy < 3 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except contraceptives)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Pregnancy, planned pregnancy or lactating
* History or family history of epilepsia

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-19 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Retinal blood-flow variation over time | 14 +/- 3 days
  as measured using DOCT

SECONDARY OUTCOMES:
Flicker induced blood flow alterations | 14 +/- 3 days
  as measured using DOCT
Flicker induced vasodilatation and hyperemia | 14 +/- 3 days
  as measured using DOCT and DVA

CONTACTS AND LOCATIONS:
Overall Officials: Doreen Schmidl, MD, PhD, Principal Investigator — Medical University of Vienna, Department of Clinical Pharmacology
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Werkmeister RM, Dragostinoff N, Palkovits S, Told R, Boltz A, Leitgeb RA, Groschl M, Garhofer G, Schmetterer L. Measurement of absolute blood flow velocity and blood flow in the human retina by dual-beam bidirectional Doppler fourier-domain optical coherence tomography. Invest Ophthalmol Vis Sci. 2012 Sep 12;53(10):6062-71. doi: 10.1167/iovs.12-9514. PMID 22893675
- [Background] Doblhoff-Dier V, Schmetterer L, Vilser W, Garhofer G, Groschl M, Leitgeb RA, Werkmeister RM. Measurement of the total retinal blood flow using dual beam Fourier-domain Doppler optical coherence tomography with orthogonal detection planes. Biomed Opt Express. 2014 Jan 28;5(2):630-42. doi: 10.1364/BOE.5.000630. eCollection 2014 Feb 1. PMID 24575355
- [Background] Werkmeister RM, Palkovits S, Told R, Groschl M, Leitgeb RA, Garhofer G, Schmetterer L. Response of retinal blood flow to systemic hyperoxia as measured with dual-beam bidirectional Doppler Fourier-domain optical coherence tomography. PLoS One. 2012;7(9):e45876. doi: 10.1371/journal.pone.0045876. Epub 2012 Sep 18. PMID 23029289
- See also: Medical University of Vienna, Department of Clinical Pharmacology — https://klpharm.meduniwien.ac.at/